CLINICAL TRIAL: NCT03613350
Title: Prevalence Rates of Urodynamic Stress Incontinence, Bladder Oversensitivity/Detrusor Overactivity or Both and Their Clinical and Urodynamic Findings in Women With ≥Stage II Cystocele
Brief Title: Prevalence Rates of USI, BO, DO and Their Clinical and Urodynamic Findings in Women With ≥Stage II Cystocele
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805024RINB
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Lower Urinary Tract Symptom in Severe Cystocele Women
Keywords: Cystocele; Urodynamic stress incontinence; Detrusor overactivity; Pad test; Urodynamic study
MeSH Terms: conditions — Cystocele; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Urodynamic stress incontinence: Urodynamic study incontinence Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20-minute pad testing and urodynamic studies in a medical center were reviewed. USI included evident USI and occult USI, which were classified according to pad weight before and after prolapse reduction.
  Interventions: Diagnostic Test: Pad test
- USI+BO/DO: Urodynamic study incontinence + bladder oversensitivity / detrusor overactivity Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20-minute pad testing and urodynamic studies in a medical center were reviewed. USI included evident USI and occult USI, which were classified according to pad weight before and after prolapse reduction.BO was defined as <300 mL of the volume at strong desire to void during filling cystometry. Detrusor overactivity was defined as evidence of spontaneous detrusor contractions occurring during bladder filling or an uninhibited detrusor contraction occurring at a cystometric capacity that usually results in voiding.
  Interventions: Diagnostic Test: Pad test
- BO/DO: Urodynamic study incontinence + bladder oversensitivity / detrusor overactivity Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20-minute pad testing and urodynamic studies in a medical center were reviewed. BO was defined as <300 mL of the volume at strong desire to void during filling cystometry. Detrusor overactivity was defined as evidence of spontaneous detrusor contractions occurring during bladder filling or an uninhibited detrusor contraction occurring at a cystometric capacity that usually results in voiding.
  Interventions: Diagnostic Test: Pad test
- No demonstrated USI+BO/DO: Urodynamic study incontinence + bladder oversensitivity / detrusor overactivity Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20-minute pad testing and urodynamic studies in a medical center were reviewed. No urodynamic stress incontinence, no bladder oversensitivity nor detrusor overactivity was noted in this group.
  Interventions: Diagnostic Test: Pad test

INTERVENTIONS:
Diagnostic Test: Pad test — 20-minutes pad test and urodynamic study (including uroflowmetry, filling and voiding cystometry, and urethral pressure profile) were conducted to every patient.
  Other Names: urodynamic study

SUMMARY:
Prevalence rates of urodynamic stress incontinence (USI), bladder oversensitivity (BO) /detrusor overactivity (DO) or both and their related clinical and urodynamic findings in women with ≥ pelvic organ prolapse quantification stage II cystocele are important for clinical consultation. Thus, the aim of this study was to elucidate the above findings and between-group associations.

DETAILED DESCRIPTION:
Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent 20-minute pad testing and urodynamic studies in a medical center were reviewed. ANOVA test and post-hoc testing with bonferroni's correction were used for statistical analysis. USI included evident USI and occult USI, which were classified according to pad weight before and after prolapse reduction. BO was defined as <300 mL of the volume at strong desire to void during filling cystometry. Those women without USI, BO or DO were allocated into the no demonstrated USI+BO/DO group.

ELIGIBILITY:
Inclusion Criteria:

1. Age >20y/o
2. Severe cystocele, ie, more than stage 2
3. Complete pad test and urodynamic study

Exclusion Criteria:

1. Pregnancy
2. Urinary tract infection
3. Had received pelvic reconstruction

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with ≥stage II cystocele.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
USI | Between November 2011 and January 2017
  Urodynamic stress incontinence was noted during examination
BO/DO | Between November 2011 and January 2017
  Bladder oversensitivity/detrusor overactivity was noted during examination

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD